CLINICAL TRIAL: NCT04009460
Title: An Open-label, Multicenter, Dose-escalation and Cohort Expansion Phase 1 Clinical Study of ES101 in Patients With Advanced Solid Tumors
Brief Title: A Study of ES101 (PD-L1x4-1BB Bispecific Antibody) in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's clinical development strategy adjustment
Sponsor: Elpiscience Biopharma, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ES101-1001; CTR20190888 (Registry Identifier: NMPA of China)
Record Dates: First submitted 2019-07-03; First posted 2019-07-05 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Solid Tumors; Neoplasms; Malignant Tumor
Keywords: ES101; solid tumor; phase 1; PD-L1; 4-1BB; INBRX-105; PD-L1×4-1BB; 41BB; PDL1
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A dose escalation (Experimental): ES101 will be escalated in patients with advanced solid tumors.
  Interventions: Drug: ES101
- Part B expansion (Experimental): Subjects with solid tumors will be treated with single-agent ES101 at either specified dose levels or RP2D.
  Interventions: Drug: ES101

INTERVENTIONS:
Drug: ES101 — ES101 is administered via intravenous infusion, once every 14 days, every 28 days as a treatment cycle.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerance and Dose-Limiting Toxicity (DLT) of recombinant humanized PD-L1/4-1BB bispecific antibody (ES101) in patients with advanced solid tumors.

DETAILED DESCRIPTION:
ES101 (INBRX-105; PDL1x4-1BB antibody) is a recombinant humanized bispecific IgG1 antibody targeting human PD-L1 and 4-1BB. This is an open-label, multicenter, dose-escalation and cohort expansion phase 1 clinical study to evaluate the safety and pharmacokinetic characteristics and preliminary anti-tumor activity of ES101 in patients with advanced malignant solid tumors whose disease has progressed despite standard therapy, or who has no further standard therapy, or who is unsuitable for available standard treatment options.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥ 18 years.
2. Subject has pathological or cytological diagnosed advanced malignant solid tumor, whose disease has progressed despite standard therapy, or who has no further standard therapy, or who is unsuitable for available standard treatment options
3. Part A: There is no mandatory requirement for PD-L1 expression status of subject's tumor tissue. Part B:Tumor tissue of subject should be PD-L1 positivity by immunohistochemistry (IHC).
4. Subjects in part A shall have at least one evaluable lesion, and subjects enrolled in part B shall have at least one measurable lesion (RECIST v1.1). Tumor lesions located in previously irradiated (or other local treated) areas will be considered measurable, provided that there has been clear imaging-based progression of the lesions since the time of radiation.
5. Adequate hematologic, coagulation, hepatic and renal function as defined per protocol.
6. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.
7. Estimated life expectancy, in the judgment of the investigator, of at least 12 weeks.
8. Male and female subjects of childbearing potential and their spouses must be willing to use feasible contraceptive methods considered effective by the investigator, from the time of signing informed consent and for the duration of study participation through 3 months, following the last dose of study drug. Postmenopausal women are considered to have no fertility potential only if menostasis lasts for at least 12 months.
9. Ability to understand and the willingness to sign a written informed consent form

Exclusion Criteria:

1. Prior exposure to 4-1BB agonists.
2. Receipt of any anticancer investigational product or any approved drug(s) or biological products (except hormone-replacement therapy, testosterone or oral contraceptives) within 4 weeks prior to the first dose of study drug. Previous exposure to oral fluorouracils or small molecular targeted drugs require a minimum washout period of 2 weeks or 5 half-lives prior to the first dose of study drug (whichever is longer). Previous exposure to mitomycin C or nitrosourea requires a minimum washout period of 6 weeks prior to the first dose of study drug.
3. Known allergies to CHO-produced antibodies, which in the opinion of the Investigator suggests an increased potential for an adverse hypersensitivity to ES101.
4. Primary or metastatic brain or meningeal tumors.
5. Patients with other malignancies previously or currently shall be excluded in Part B.
6. Grade ≥ 3 immune-related adverse events (irAEs) or irAE that lead to discontinuation of prior immunotherapy. Some exceptions as defined per protocol apply.
7. Active autoimmune disease or documented history of autoimmune disease that required systemic steroids or other immunosuppressive medications. Certain exceptions as defined in protocol apply.
8. Treatment with systemic immunosuppressive medications within 4 weeks prior to the first dose of study drug. Certain exceptions as defined in protocol apply.
9. Active interstitial lung disease (ILD) or pneumonitis or a history of ILD or pneumonitis requiring treatment with steroids or immunosuppressive medications..
10. Subjects who received G-CSF, GM-CSF, Thrombopoietic drugs or EPO within 14 days prior to the first dose of the study drug.
11. Any evidence of hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection.
12. History of hepatitis (non-alcohol steatohepatitis, alcohol or drug-related, autoimmune) or cirrhosis.
13. Clinically significant cardiac condition.
14. History of pulmonary embolism within 12 weeks prior to the first dose of study drug.
15. Major surgery within 4 weeks prior to enrollment on this trial.
16. Systemic anti-infectious drug treatments within 4 weeks prior to the first dose of study drug.
17. Prior organ allograft transplantations or allogeneic peripheral blood stem cell (PBSC) or bone marrow (BM) transplantation.
18. Live viral vaccine therapies within 4 weeks prior to the first dose of study drug.
19. Subject has not recovered from all AEs of previous anticancer therapies to baseline or ≤ Grade 1 per CTCAE v5.0 before teh first dose of study drug. Certain exceptions as defined in protocol apply.
20. Pregnant or nursing females.
21. Any known, documented, or suspected history of substance abuse that would preclude subject from participation, unless clinically justified (i.e., will not interfere with study participation and/or will not compromise trial objectives) per judgment of the Investigator and with approval of the Medical Monitor or Study Director.
22. The subject is inappropriate to participate in this study for other reasons in the judgment of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of of ES101 | Up to 2-3 years
  The MTD and/or RP2D of ES101 will be determined.
Frequency of adverse events of ES101 | Up to 2-3 years
  Adverse events will be assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Severity of adverse events of ES101 | Up to 2-3 years
  Severity of adverse events will be assessed and assigned by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.

SECONDARY OUTCOMES:
Area under the serum concentration time curve (AUC) of ES101 | Up to 2-3 years
  Area under the serum concentration time curve (AUC) of ES101 will be determined.
Maximum observed serum concentration (Cmax) of ES101 | Up to 2-3 years
  Maximum observed serum concentration (Cmax) of ES101 will be determined.
Trough observed serum concentration (Ctrough) of ES101 | Up to 2-3 years
  Trough observed serum concentration (Cmax) of ES101 will be determined.
Time to Cmax (Tmax) of ES101 | Up to 2-3 years
  Time to Cmax (Tmax) of ES101 will be determined.
Immunogenicity of ES101 | Up to 2-3 years
  Frequency of anti-drug antibodies (ADA) against ES101 will be determined.
Anti-tumor activity of ES101 | Up to 2-3 years
  Tumor response will be determined by the revised Response Evaluation Criteria in Solid Tumors version 1.1 (RECISTv1.1).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No